CLINICAL TRIAL: NCT02635958
Title: Validation of the InBody 770® for the Assessment of Body Composition
Brief Title: InBody Validation Study
Acronym: InBody
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: BioSpace, Inc. (Industry)
Responsible Party: Principal Investigator, Ryan T. Hurt, M.D., Ph.D., PI, Mayo Clinic
Other Study IDs: 14-004659
Record Dates: First submitted 2015-12-17; First posted 2015-12-21 (Estimated); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Validation Study
Keywords: Body Mass Index; BMI; InBody; iDXA; validation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Group 1: BMI 18.5 to 24.9
- Group 2: BMI 25 to 29.9
- Group 3: BMI 30 to 34.9
- Group 4: BMI ≥ 35

SUMMARY:
With, one in three Americans now having a body mass index (BMI) greater than 30, and the fastest growing segment of the population having a BMI greater than 40, it is paramount to conduct validation of approaches to measure body composition. Currently the dual-energy x-ray absorptiometry (iDXA) is the gold standard for measuring the body composition. But it is often difficult to perform since it is limited to specific height, weight and BMI's. InBody is a tool which uses bio electric impedance to measure the body composition. This study will compare both approaches. Validation is necessary as it is clinically quite pertinent to accurately assess a patients' body fat percentage, fat free mass, and total body water and changes that are occurring with nutritional support.

DETAILED DESCRIPTION:
This study will use a stratified design. Eligible participants will be categorized with BMI category to receive InBody followed by iDXA. A total of 176 participants will be placed in 1 of 4 arms (n = 44 per arm) based on their BMI: 1) 18.5-24.9; 2) 25-29.9; 3) 30-34.9; and 4) ≥ 35. Within these arms, the 44 participants will participate in an InBody 770® body composition measure as well as an iDXA body composition measure.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years of age
* Have a Body Mass Index ≥ 18.5 kg/m2

Exclusion Criteria:

* Are not English speaking
* Are younger than 18 years of age
* Weigh more than 450 lbs
* Taller than 6'6" due to size constraints of the iDXA
* Have a pacemaker, defibrillator, artificial lung, artificial heart, electrocardiograph, or nerve simulator
* People having radioactive iodine thyroid treatment.
* People who have had a nuclear medicine study or a barium X-ray within the last 5 days.
* People with large amounts of metal in their bodies.
* People with arthritis of the spine recorded in the medical record.
* Are pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with a BMI greater than 18.5 and weigh no more than 450 lbs.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Body Composition Measures | 1 day
  compare body composition measures between InBody and iDXA

CONTACTS AND LOCATIONS:
Overall Officials: Ryan T Hurt, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials